CLINICAL TRIAL: NCT05304377
Title: A Phase 1a/1b Study of ELVN-001 for the Treatment of Chronic Myeloid Leukemia
Brief Title: A Phase 1a/1b Study of ELVN-001 for the Treatment Chronic Myeloid Leukemia
Acronym: CML
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Enliven Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ELVN-001-101
Record Dates: First submitted 2022-03-15; First posted 2022-03-31 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Chronic Myeloid Leukemia; Chronic Phase Chronic Myeloid Leukemia, BCR-ABL1 Positive; Cml
Keywords: CML; Tyrosine kinase inhibitor; T315I; T315I mutant; BCR-ABL; ENABLE; active site inhibitor of BCR-ABL
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1a Dose Escalation (Experimental): ELVN-001 administered in 3+3 dose escalation
  Interventions: Drug: ELVN-001
- Phase 1b Dose Expansion (non-T315I) (Experimental): ELVN-001 administered at one or more recommended dose(s) for expansion in CML without T315I mutations
  Interventions: Drug: ELVN-001
- Phase 1b expansion (T315I) (Experimental): ELVN-001 administered at the recommended dose for expansion for CML with T315I mutation
  Interventions: Drug: ELVN-001

INTERVENTIONS:
Drug: ELVN-001 — orally once or twice daily

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and determine the recommended dose for further clinical evaluation of ELVN-001 in patients with chronic myeloid leukemia with and without T315I mutations in patients who are relapsed, refractory or intolerant to TKIs.

DETAILED DESCRIPTION:
This first-in-human trial with ELVN-001 is a dose escalation study with the primary purpose to identify the recommended dose(s) for expansion (RDEs) of single agent ELVN-001 in chronic phase CML with or without T315I mutations. The safety, tolerability and pharmacokinetic profile of ELVN-001 will be assessed together with an evaluation of changes in BCR-ABL1 transcript. An understanding of the safety profile, PK and preliminary evidence of anti-CML activity will be used to inform future development of ELVN-001 in adults with CML. By virtue of its predicted pharmacological profile ELVN-001 has the potential to be tolerable and achieve a deep molecular response in patients with CML with or without T315I mutations who do not tolerate or benefit from available TKIs.

ELIGIBILITY:
Inclusion Criteria:

* BCR-ABL1 positive CML in chronic phase, with or without T315I mutation.
* US: The patient has failed or is intolerant to at least one prior second-generation tyrosine kinase inhibitor (TKI) or asciminib. Rest of World: The patient has failed, is intolerant to, or not a candidate for, available therapies known to be active for treatment of their CML (country-specific criteria may vary).
* ECOG performance status of 0 to 2.
* Adequate hematologic, hepatic and renal function.
* Prior bone marrow transplant allowed if ≥ 6 months prior to the first dose of ELVN-001.

Exclusion Criteria:

* Treatment with anti-cancer or anti-CML therapy within 7 days or 5 half-lives, whichever is longer.
* History of acute tyrosine kinase inhibitor (TKI)-related pancreatitis within 6 months of study entry. Active chronic pancreatitis, or pancreatic disease due to any cause.
* QTc >470 ms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-05-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Incidence of dose limiting toxicities | 28 days
  DLTs will be used to support that the recommended doses for expansion are </= MTD
Phase 1a: Incidence of adverse events (AEs) | up to 28 days
  Adverse events will be used to support that the recommended doses for expansion are likely to be tolerable
Phase 1a: Incidence of clinically significant laboratory abnormalities | up to 28 days
  Clinically significant laboratory abnormalities will be used to support that the recommended doses for expansion are likely to be tolerable
Phase 1a: Incidence of clinically significant ECG abnormalities | up to 28 days
  Clinically significant ECG abnormalities will be used to support that the recommended doses for expansion are likely to be tolerable
Phase 1b: Incidence of adverse events | up to 3 years
  Adverse events will be used to support that the dose(s) evaluated in expansion is tolerable
Phase 1b: Incidence of clinically significant laboratory abnormalities | up to 3 years
  Clinically significant ECG abnormalities will be used to support that the dose(s) evaluated in expansion is tolerable
Phase 1b: Incidence of clinically significant ECG abnormalities | up to 3 years
  Clinically significant ECG abnormalities will be used to support that the recommended dose(s) evaluated in expansion is tolerable

SECONDARY OUTCOMES:
Phase 1a and 1b: area under the curve | 6 months
  PK parameter based on measurement of drug concentration in blood over time
Phase 1a and 1b: maximum concentration | 6 months
  PK parameter based on measurement of drug concentration in blood
Phase 1a and 1b: time of maximum concentration | 6 months
  PK parameter which is the time at which the highest concentration of drug in the blood is measured
Phase 1a and 1b: minimum concentration | 6 months
  PK parameter based on the measurement of the drug concentration that is at the lowest level once steady state has been achieved.
Phase 1a and 1b: Molecular response (MR) | up to 3 years
  measured by quantitative polymerase chain reaction of BCR-ABL transcript levels
Phase 1b: Duration of Molecular Response | up to 3 years
  Time from first molecular response (as measured by quantitative polymerase chain reaction of BCR-ABL transcript levels) to loss of response or discontinuation of study drug
Phase 1b: Complete Hematologic Response (CHR) | up to 3 years
  The proportion of patients who achieve a CHR who are not in CHR at baseline

CONTACTS AND LOCATIONS:
Locations (46):
- United States (4):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Oregon Health & Science University-Knight Cardiovascular Institute, Portland, Oregon
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Royal Adelaide Hospital, Adelaide, Australia
- Belgium (3):
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - CHU Liege, Liège
- University Health Network (UHN) - Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- France (7):
  - CHU Amiens Picardie Site Sud, Amiens
  - Institut Bergonie - Centre Regional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux
  - Centre Hospitalier de Versailles (CHV), Le Chesnay
  - CHRU de Lille - Hopital Calmette-Boulevard du Pr Leclercq CHRU Lille, Lille
  - Centre Hospitalier Universitaire (CHU) De Limoges Hopital Dupuytren, Limoges
  - Centre Leon Berard, Lyon
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
- Germany (7):
  - Uniklinik RWTH Aachen Medizinische, Aachen
  - Charite Campus Virchow, Berlin
  - Klinikum der Goethe Universitat, Frankfurt
  - Universitaetsklinikum Des Saarlandes Und Medizinische Fakultaet Der Universitaet Des Saarlandes, Homburg
  - Universitaetsklinikum Jena, Jena
  - Medizinische Universitatsklinik Mannheim der Universitat Heidelberg, Mannheim
  - Universitaetsmedizin Rostock, Rostock
- Hungary (2):
  - Semmelweis Egyetem, Belgyogyaszati es Onkologiai Klinika, Budapest
  - Pecsi Tudomanyegyetem Klinikai Kozpont (University of Pecs, Clinical Centre), Pécs
- Israel (3):
  - Hadassah Medical Center, Jerusalem
  - The Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
- Azienda Ospedaliero Universitaria Delle Marche, Ancona, Italy
- Radboud University Medical Center, Nijmegen, Netherlands
- Poland (3):
  - Szpital Specjalistycnzy im. Jedrzeja Sniadeckiego w Nowym Saczu, Nowy Sącz
  - MICS Centrum Medyczne Torun, Torun
  - Instytut Hematologii I Transfuzjologii, Warsaw
- South Korea (5):
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Keimyung University Dongsan Hospital, Daegu
  - Uijeongbu Eulji Medical Center, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun
  - Samsung Medical Center, Seoul
- Spain (5):
  - Hospital Del Mar, Barcelona
  - Hospital Universitario de Gran Canaria Dr. Negrin, Servicio Canario e Salud (SCS), Las Palmas de Gran Canaria
  - Hospital Universitario La Paz, Madrid
  - Complejo Hospitalario de Toledo - Hospital Virgen de la Salud, Toledo
  - Universitat de Valencia - Hospital Universitari i Politecnic La Fe de Valencia (Hospital La Fe Bulevar Sur), Valencia
- United Kingdom (3):
  - Beatson West of Scotland Cancer Centre, Gartnavel General Hospital, Glasgow
  - Hammersmith Hospital Imperial College Healthcare NHS Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No